CLINICAL TRIAL: NCT02848261
Title: Remote Monitoring of Diabetes in Young Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Colorado, Denver (Other); Indiana University (Other); University of South Florida (Other)
Responsible Party: Principal Investigator, Korey Hood, Professor, Stanford University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 37360
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Developmental Demands (Experimental): Provide education on using diabetes technology in various settings and formats in this age group, and increase ability for real-time problem-solving.
  Interventions: Behavioral: Developmental Demands
- Distress Reduction (Experimental): Identify and reduce parent distress symptoms and worries. Provide strategies for obtaining social support.
  Interventions: Behavioral: Distress Reduction
- Remote Monitoring (Experimental): Optimize the use of remote monitoring by focusing on situational demands and problem solving.
  Interventions: Behavioral: Remote Monitoring
- Fear of Hypoglycemia (Experimental): Decrease fear of hypoglycemia, particularly focusing on overnight glycemic control.
  Interventions: Behavioral: Fear of Hypoglycemia
- No Intervention (Placebo Comparator): Serves as the control group comparator. No intervention provided.
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: Developmental Demands — Education and training related to use of CGM in this age group
  Arms: Developmental Demands
Behavioral: Distress Reduction — Education and training on reducing distress
  Arms: Distress Reduction
Behavioral: Remote Monitoring — Education and training on the use of remote monitoring
  Arms: Remote Monitoring
Behavioral: Fear of Hypoglycemia — Education and training on reducing fear of hypoglycemia
  Arms: Fear of Hypoglycemia
Behavioral: No intervention — No intervention - serves as the control group
  Arms: No Intervention

SUMMARY:
The primary objective of this project is to examine the impact of a continuous glucose monitoring (CGM) intervention on health and psychological outcomes in young children with type 1 diabetes (T1D).

ELIGIBILITY:
To be eligible for the study, a child must meet the following criteria:

1. Diagnosis of type 1 diabetes according to American Diabetes Association diagnostic criteria
2. Time since diagnosis of at least six months
3. Age between 2 and 6 years at enrollment
4. Parental consent to participate in the study
5. No severe medical conditions, which in the opinion of the investigators are likely to hinder participation in this clinical trial.
6. If current use of CGM, A1c has to be above 7.5%; value obtained within 3 months of enrollment
7. Own and use an iPhone, or be willing/able to carry a study-supplied wi-fi enabled iPod

To be eligible for the study, a parent must meet the following criteria:

1. Parent or legal guardian of a child with type 1 diabetes meeting the "child" criteria outlined above
2. Age of 18.0 years or older
3. Parent comprehends written English
4. Parent understands the study protocol and signs the informed consent document
5. Parent has access to a personal computer to upload diabetes devices and send to research team

The presence of any of the following is an exclusion for the study:

1. Child has a medical disorder that in the judgment of the investigator will interfere with completion of any aspect of the protocol (e.g., pregnancy, kidney disease, adrenal insufficiency, skin condition that may hinder sensor application).
2. Child has a neurologic disorder that in the judgment of the investigator will affect completion of the protocol
3. Current use of oral glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
4. Child is unable to completely avoid acetaminophen for duration of study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Time spent in blood glucose range | Change over 6 months
  Increasingly it is recognized that the percent time spent in a target blood glucose range, which is set by the American Diabetes Association, is an important outcome. This measure will be used as a primary outcome and derived from objective data downloads.
Pediatric Quality of Life Inventory | Change over 6 months
  This is a measure of health-related quality of life. It is used to understand the broader impact on quality of life which includes social, psychological, and health aspects of daily living.

SECONDARY OUTCOMES:
A1c | Change over 6 months
  The hemoglobin A1c value is a biologic measure of the glycemia that is the gold standard measure of "control" of diabetes. Collected through a blood sample.
Problem Areas in Diabetes | Change over 6 months
  This measure captures areas that are reported as problems for people with diabetes. Participants in the study report on daily problems with diabetes via this measure.
Diabetes Distress Scale | Change over 6 months
  This measure is widely used to capture the psychological distress experienced in relation to diabetes.
Patient Health Questionnaire 9 | Change over 6 months
  This is a widely used measure that captures depressive symptoms. It is reported by the participants.
State-Trait Anxiety Inventory | Change over 6 months
  This is a widely used measure of anxiety symptoms. It is reported by the participant.
Pittsburgh Sleep Quality Index | Change over 6 months
  This questionnaire measures the degree to which sleep is disrupted and the quality of sleep experienced by participants.
Hypoglycemic Fear Survey | Change over 6 months
  People with diabetes worry about hypoglycemia. This measure captures those worries and is reported by participants.
Hypoglycemic Confidence Questionnaire | Change over 6 months
  Hypoglycemia needs to be managed in various daily situations. This questionnaire captures confidence of the participants in those various situations.
Glucose Monitoring System Satisfaction Survey | Change over 6 months
  This a measure used to capture overall satisfaction with glucose monitoring devices used by participants.
General and diabetes-specific technology use | Change over 6 months
  This measure has questions on attitudes and use of various general technologies (e.g., smartphone) and diabetes devices.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University; Kimberly Driscoll, PhD, Principal Investigator — University of Colorado, Denver; Linda DiMeglio, MD, Principal Investigator — Indiana University; Henry Rodriguez, MD, Principal Investigator — University of South Florida
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - Indiana University, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes